CLINICAL TRIAL: NCT05279612
Title: Effect Analysis of Neoadjuvant Chemoradiotherapy Combined With Radical Surgery ( CME + D3 ) for Advanced Colon Cancer : Prospective, a Single-arm, Single Central, Clinical Trial Research
Brief Title: Effect Analysis of Neoadjuvant Chemoradiotherapy Combined With Surgery in Laparoscope for Advanced Colon Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: K202012-12
Record Dates: First submitted 2021-02-06; First posted 2022-03-15 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Colon Neoplasm
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- neoadjuvant chemoradiotherapy group: preoperative 1 circle chemotherapy(CapeOX) combined with short-course radiotherapy ，Surgical treatment(CME+D3) after four weeks of 2 circle chemotherapy(CapeOX).
  Interventions: Radiation: Short-term neoadjuvant chemoradiotherapy
- neadjuvant chemotherapy group: preoperative 3 circle chemotherapy(CapeOX) combined with surgical treatment(CME+D3)

INTERVENTIONS:
Radiation: Short-term neoadjuvant chemoradiotherapy — Short-term radiotherapy ( 25 Gy, 5f ) + XELOX regimen was performed before operation for two cycles. After the condition was evaluated by enhanced CT, whether the patients belonged to PD, SD, PR and CR was analyzed (reference RECIST 1.1). Surgery was performed four weeks after chemotherapy.
  Groups: neoadjuvant chemoradiotherapy group

SUMMARY:
In this study, a randomized controlled trial was conducted on advanced colon cancer patients with preoperative tumor staging T1-4/N1-2/M0 or T4/N0/M0 to determine the effectiveness of preoperative short-term radiotherapy combined with chemotherapy and whether it can effectively reduce the postoperative local recurrence rate, so as to provide better treatment for colon cancer patients and improve the oncological treatment effect of colon cancer.

DETAILED DESCRIPTION:
This is prospective,a single-arm, single center, clinical trail study.The patient entered the study after meeting that criteria.The ORR, R0 resection, OS and DFS of patients and neoplasm down-staging status,etc would be compared.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of colon neoplasm
* 18 years to 70 years
* Preoperative abdominal enhanced CT or MRI showed cT4, cN0-2
* ECOGS score≤2
* thoraco-abdomina CT showed no obvious metastasis（The CT of liver and lung show uncertainty tubercle,suggestive performed PET-CT) cT4,cN0-2,M0 radiography Inclusion Criteria（according postoperative enhanced CT or MRI）
* progress tubercle penetrate peritoneotome base
* progress tubercle penetrate serous surface of neighboring organ
* progress tubercle development by late mesentery or side abdominis

Exclusion Criteria:

* Appeared other system cancer
* Patient with postoperative recurrent of colon cancer
* Patient with malignancies history in recent 5 years
* Pregnant or female of suckle period
* The patient have adjuvant radiotherapy record in other system cancer before this time treatment，and Patient with surgical contraindications.
* The patient have accepted adjuvant chemoradiotherapy before this time treatment.
* Distant metastasis found during surgery
* Patients with poor radiotherapy compliance and difficulty in coordination
* Patients with mental disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosis of colon neoplasm, 18 years to 70 years, Preoperative abdominal enhanced CT or MRI showed cT4, cN0-2, thoraco-abdomina CT showed no obvious metastasis（The CT of liver and lung show uncertainty tubercle,suggestive performed PET-CT), cT4,cN0-2,M0 radiography Inclusion Criteria（according postoperative enhanced CT or MRI）
Sampling Method: Non-Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Investigate patients ORR | 7 days after surgery
  Investigate patients ORR(objective response rate ) include CR(complete response) and PR(partial response)

SECONDARY OUTCOMES:
neoplasm down-staging status | one month after surgery
  Observation of neoplasm down-staging status in patients according to RECIST 1.1
Investigate operation safety score | one month after surgery
  Operation safety reference Clavien degree of postoperative complication
local recurrent rate of neoplasm | 2 years after surgery
  Observation local recurrent rate of neoplasm in patients
Quality of life score | one month after surgery
  Investigate postoperative Quality of life in patients after surgery
Investigate patience pRR (pathologic response rate) | 7 days after surgery
  According to the English version of the Japanese Gastric Cancer Classification (JCGC) 3rd edition, pRR is defined as survival of tumor cells remaining in less than 2/3 of the tumor area (level Ib or higher)
R0 resection | immediately after surgery
  R0 resection indicates a microscopically margin-negative resection,in which no gross or microscopic tumor remains in the primary tumor bed

CONTACTS AND LOCATIONS:
Overall Officials: Nan Wang, Doctor, Study Director — General Surgery,Tang-Du of Military Medical University
Locations (1):
- General Surgery Gastrointestinal Department,Tang-Du of Fourth Military Medical University, Xi’an, Shanxi, China